CLINICAL TRIAL: NCT01811043
Title: Improving Biopsy Experiences Study for Women
Acronym: IBEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00038873
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2017-11

CONDITIONS: Imaging Guided Breast Biopsy
Keywords: breast biopsy; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Guided Meditation (Experimental): Guided meditation is played via headphones during biopsy
  Interventions: Behavioral: Guided Meditation
- Music (Active Comparator): Music is played via headphones during biopsy
  Interventions: Behavioral: Music
- Supportive Dialogue (Placebo Comparator): Supportive dialogue is provided during biopsy by the radiologist performing the procedure
  Interventions: Behavioral: Supportive Dialogue

INTERVENTIONS:
Behavioral: Guided Meditation
  Arms: Guided Meditation
Behavioral: Music
  Arms: Music
Behavioral: Supportive Dialogue
  Arms: Supportive Dialogue

SUMMARY:
The goal of this study is to examine whether a guided meditation intervention will reduce anxiety and distress as compared to a music intervention or radiologist supportive dialogue in women undergoing imaging-guided core needle breast biopsies. Both the guided meditation and music interventions are administered through use of headphones during routine outpatient imaging-guided core needle breast biopsies. Women in the guided meditation and music conditions will be given a CD with instructions for home practice. Women complete follow-up questionnaires in the 12 months after biopsy. Receipt of recommended follow-up care is examined for 60 months.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Undergoing imaging guided core needle biopsy
* Mammography or ultrasound Breast Imaging - Reporting and Data System(BI-RADS) final assessment category 3,4a-c, or 5
* Able to speak and read English
* Able to provide meaningful consent

Exclusion Criteria:

* significant hearing impairment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety | Change in anxiety from baseline (i.e., pre biopsy) assessment to post biopsy assessment will be examined. Participants will be followed for the duration of the biopsy, with an expected average of 1.5 hours between assessments.
  Anxiety is measured using the State Anxiety Scale of the State Trait Anxiety Inventory. Women complete this self-report measure at baseline (i.e., immediately prior to biopsy in the biopsy clinic) and immediately post-biopsy. Change in anxiety will be measured as change from baseline to post biopsy (i.e., post biopsy anxiety - baseline anxiety.) The expected duration from baseline to post biopsy assessment is expected to be an average of 1.5 hours.

SECONDARY OUTCOMES:
Rates of adherence to recommended follow-up care | 60 months following biopsy
  Adherence to recommended mammography and clinical breast exam will be assessed for 60 months following biopsy. Adherence (i.e., repeated on schedule mammograms; repeated on schedule clinical breast exams) at 60 months post biopsy will be compared across study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Scott Soo, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States